CLINICAL TRIAL: NCT00927992
Title: Liver Transplantation in Haemophilia Patients in Spain
Brief Title: Study Evaluating Liver Transplantation in Haemophilia Patients in Spain
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1831011; 3082B1-4436 (Other: Wyeth)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Hemophilia; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with haemophilia who undergo liver transplantation: Patients with haemophilia who underwent liver transplantation and who have been followed up at any site in Spain.
  Interventions: Other: Epidemiological Non interventional

INTERVENTIONS:
Other: Epidemiological Non interventional — Epidemiological Non interventional

SUMMARY:
This study will analyze survival and outcome of patients with severe haemophilia who undergo liver transplantation in Spain

DETAILED DESCRIPTION:
Probability Sample

ELIGIBILITY:
Inclusion Criteria:

* Patients with haemophilia who underwent liver transplantation and who have been followed-up at any site in Spain.

Exclusion Criteria:

* Patients without informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia who underwent liver transplantation and who have been followed-up at any site in Spain.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B1-4436&StudyName=Study%20Evaluating%20Liver%20Transplantation%20in%20Haemophilia%20Patients%20in%20Spain%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemophiliac Participants With Liver Transplant: Participants with hemophilia (type A or B) who had undergone a liver transplant were observed for 3 months.
Period: Overall Study
Arm/Group | Hemophiliac Participants With Liver Transplant
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 45.45 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Number of participants with Type A and B Hemophilia [Number; unit: participants]
  Type A | 9
  Type B | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Immunosuppressive Therapy After Liver Transplantation
Description: Cyclosporine, corticosteroids, tacrolimus, mycophenolate mofetil, everolimus were considered as immunosuppressive therapy after liver transplantation.
Time Frame: Post liver transplantation up to Month 3
Population: Evaluable population included all the participants who met the eligibility criteria.
Measure: Number; unit: Participants
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 11
Participants
  Cyclosporine | 7
  Corticosteroids | 6
  Tacrolimus | 4
  Mycophenolate Mofetil | 3
  Everolimus | 1

2. Primary Outcome: Number of Participants With Acute Rejection of Liver Transplant
Description: Any acute rejection of the liver transplant was clinically suspected and biopsy proven by central pathologist.
Time Frame: Post liver transplantation up to Month 3
Population: Evaluable population included all the participants who met the eligibility criteria.
Measure: Number; unit: Participants
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 11
Participants | 0

3. Primary Outcome: Number of Participants With Hepatitis C Viral Infection Recurrence After Liver Transplantation
Description: Number of participants who had liver transplantation after cirrhosis due to hepatitis C virus (HCV) infection and experienced recurrence of HCV infection post liver transplantation.
Time Frame: Post liver transplantation up to Month 3
Population: Evaluable population included all the participants who met the eligibility criteria.
Measure: Number; unit: Participants
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 11
Participants | 4

4. Primary Outcome: Number of Participants Who Survived After Liver Transplantation
Description: Number of participants who survived after liver transplantation was reported. The death reported was a result of acute-related transplantation complications and end-stage liver disease.
Time Frame: Post liver transplantation up to Month 3
Population: Evaluable population included all the participants who met the eligibility criteria.
Measure: Number; unit: Participants
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 11
Participants | 10

5. Secondary Outcome: Number of Participants Requiring Exogenous Clotting Factor Infusion During Liver Transplantation
Description: Exogenous clotting factors administered post liver transplant included Prothromplex; platelets, fibrinogen and fresh frozen plasma (FFP) combination; FFP and platelets combination. Clotting factors were administered either as bolus or as continuous infusion.
Time Frame: Up to Day 5 post liver transplantation
Population: Evaluable population included all the participants who met the eligibility criteria.
Measure: Number; unit: Participants
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 11
Participants
  Bolus | 5
  Continuous infusion | 3

6. Secondary Outcome: Dose of Exogenous Clotting Factors Used During Liver Transplantation
Description: as for outcome 5
Time Frame: Up to Day 5 post liver transplantation
Population: Evaluable population included all the participants who met the eligibility criteria.
Measure: Mean (Standard Deviation); unit: International Unit/kilogram (IU/kg)
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 11
International Unit/kilogram (IU/kg) | 62.88 (30.09)

7. Secondary Outcome: Number of Participants With and Without Hemophilia Requiring Immunosuppressive Therapy, Had Acute Rejection, Hepatitis C Viral Infection Recurrence and Who Survived After Liver Transplantation
Time Frame: Post liver transplantation up to Month 3
Population: Data was not analyzed as only hemophiliac participants were enrolled in the study.
Arm/Group | Hemophiliac Participants With Liver Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: There were no adverse events collected in this retrospective study.
Arm/Group | Hemophiliac Participants With Liver Transplant
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No outcomes were specified in the study protocol. Designation of outcomes as primary and secondary was based on study team's input as study neither specifies nor prioritizes the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.